CLINICAL TRIAL: NCT01111487
Title: Inspiratory Muscle Recruitment in COPD Patients With the Use of Expiratory Positive Airways Pressure
Brief Title: Activity of Inspiratory Muscles With the Use of Positive Pressure in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Dannuey Machado Cardoso, Post graduation, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-500
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Electromyography; Inspiratory muscles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Active Comparator): This group will use a pressure level of 10 cmH2O.
  Interventions: Device: Expiratory positive airway pressure (EPAP) by face mask.
- Group II (Active Comparator): This group will use a pressure level of 15 cmH2O.
  Interventions: Device: Expiratory positive airway pressure (EPAP) by face mask.

INTERVENTIONS:
Device: Expiratory positive airway pressure (EPAP) by face mask. — Implementation of the EPAP as group pressure, 10 or 15 cmH2O, for 20 minutes then evaluated the electromyographic activity of muscles and sternocleidomastoid parasternal the tenth and twentieth minutes of your application.
  Other Names: PEP-mask

SUMMARY:
The objective is to evaluate whether the use of expiratory positive airway pressure (EPAP) reduces the electrical activity of the sternocleidomastoid muscle and enhances the action of the muscle in the patient parasternal ported from Chronic Obstructive Pulmonary Disease. Noting also, if the set pressure level (10 or 15 cmH2O) affects this relationship.

DETAILED DESCRIPTION:
The chronic obstructive pulmonary disease (COPD) is characterized by chronic obstruction to airflow, which leads to respiratory muscle overload and greater activation of accessory muscles of respiration, especially those active in the inspiratory phase. It is believed that the positive expiratory pressure (EPAP) reduces respiratory work, producing less activation of these muscles. Thus, we evaluate the behavior of the electrical activity of inspiratory muscles of COPD patients in response to application of expiratory positive airway pressure (EPAP), and to observe the influence of pressure level in inspiratory muscle recruitment. This will be implemented for a clinical single blinded trial (blinded to gauge the outcome) developed in the Department of Pneumology, Hospital de Clinicas de Porto Alegre (HCPA). Will be evaluated in COPD patients with a clinical diagnosis of pathology, and of both genders and should be aged between 40 and 70 years. In a first day will be collected anthropometric data, performed the lung function test for the staging of pathology and muscle strength testing. These same individuals will return to evaluate the electromyographic activity of sternocleidomastoid (SCM), and parasternal, both from the right hemisphere. This evaluation will consist in the measurement during breathing at rest (control), with the implementation of EPAP mask 10 or 15 cmH2O (state intervention) and 10 minutes after its removal. To test the lung function will be assessed using a spirometer and the lung capacity compared to the predicted in literature. As the electrical activity of muscle, will be observed the percentage of activation obtained for the highest activity (% RMS). Thus, it is expected that the implementation of EPAP promotes reduction of the electrical activity of muscle ECM and leverage the action of the parasternal muscle, affected by dynamic hyperinflation. It is also hoped that the use of blood pressure level of 15 cmH2O, compared to 10 cmH2O, the leverage effect of EPAP on the muscles of interest. The surface electromyographic evaluation is a method of relatively inexpensive and noninvasive, and is effective in evaluating the electrical potential that lies on the muscle membrane. So, will describe the effect of EPAP on the inspiratory muscles, which will be important to guide treatment of COPD patients using positive airway pressure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD in stage II or III according to classification of the Global Initiative for Chronic Obstructive Lung Disease (GOLD);
* Signing the consent form;
* Stability of clinical pathology, with no signs of exacerbation in the 30 (thirty) days prior to the inclusion in the study.

Exclusion Criteria:

* Individuals would use artificial airway;
* Hemodynamic instability;
* Body mass index (BMI) above the values considered as obese (> 30Kg/m2).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity of muscles and sternocleidomastoid parasternal | 20 minutes
  An average baseline, before the use of expiratory positive airway pressure (EPAP) to be compared with two-mediated during the 20 minutes of application of EPAP and 10 minutes after its removal.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio S Menna Barreto, Dr, Principal Investigator — Hospital of Clinicas of Porto Alegre
Locations (3):
- Brazil (3):
  - HCPA - Hospital of Clinicas of Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - University of Santa Cruz do Sul, Santa Cruz do Sul, Rio Grande do Sul

REFERENCES:
- [Background] Legrand A, Majcher M, Joly E, Bonaert A, Gevenois PA. Neuromechanical matching of drive in the scalene muscle of the anesthetized rabbit. J Appl Physiol (1985). 2009 Sep;107(3):741-8. doi: 10.1152/japplphysiol.91320.2008. Epub 2009 Jul 16. PMID 19608926
- [Background] Yokoba M, Abe T, Katagiri M, Tomita T, Easton PA. Respiratory muscle electromyogram and mouth pressure during isometric contraction. Respir Physiol Neurobiol. 2003 Aug 14;137(1):51-60. doi: 10.1016/s1569-9048(03)00092-2. PMID 12871677
- [Result] Yan S, Kaminski D, Sliwinski P. Inspiratory muscle mechanics of patients with chronic obstructive pulmonary disease during incremental exercise. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):807-13. doi: 10.1164/ajrccm.156.3.9702104. PMID 9309997
- [Result] Hudson AL, Gandevia SC, Butler JE. The effect of lung volume on the co-ordinated recruitment of scalene and sternomastoid muscles in humans. J Physiol. 2007 Oct 1;584(Pt 1):261-70. doi: 10.1113/jphysiol.2007.137240. Epub 2007 Aug 9. PMID 17690147
- [Result] CAMPBELL EJ. The role of the scalene and sternomastoid muscles in breathing in normal subjects; an electromyographic study. J Anat. 1955 Jul;89(3):378-86. No abstract available. PMID 13251968
- [Result] Levine S, Nguyen T, Friscia M, Zhu J, Szeto W, Kucharczuk JC, Tikunov BA, Rubinstein NA, Kaiser LR, Shrager JB. Parasternal intercostal muscle remodeling in severe chronic obstructive pulmonary disease. J Appl Physiol (1985). 2006 Nov;101(5):1297-302. doi: 10.1152/japplphysiol.01607.2005. Epub 2006 Jun 15. PMID 16777998
- [Result] Lien TC, Wang JH, Chang MT, Kuo CD. Comparison of BiPAP nasal ventilation and ventilation via iron lung in severe stable COPD. Chest. 1993 Aug;104(2):460-6. doi: 10.1378/chest.104.2.460. PMID 8339634
- [Result] van der Schans CP, de Jong W, de Vries G, Kaan WA, Postma DS, Koeter GH, van der Mark TW. Effects of positive expiratory pressure breathing during exercise in patients with COPD. Chest. 1994 Mar;105(3):782-9. doi: 10.1378/chest.105.3.782. PMID 8131541